CLINICAL TRIAL: NCT02459626
Title: Comparison of Non-invasive Assessment of Cardiac Fibrosis by MRI Derived T1-Mapping and Ventricular Intrinsic Diastolic Function by Pressure-volume-analysis in Patients With Heart Failure With Preserved Ejection Fraction
Brief Title: Left Ventricular Stiffness vs. Fibrosis Quantification by T1 Mapping in Heart Failure With Preserved Ejection Fraction
Acronym: STIFFMAP
Status: Completed | Type: Observational
Sponsor: Heart Center Leipzig - University Hospital (Other)
Responsible Party: Principal Investigator, Philipp Lurz, Clinical Investigator, Professor, Managing Senior Physician, Heart Center Leipzig - University Hospital
Other Study IDs: 1.02
Record Dates: First submitted 2015-05-19; First posted 2015-06-02 (Estimated); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Heart Failure With Normal Ejection Fraction
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- HFpEF and servere diastolic dysfuntion: Left ventricular ejection fraction (LV-EF) > 50%, echocardiographic criteria for diastolic dysfunction, New York Heart Association classification (NYHA)=>2, Diagnostic P-V-loops and MRI
  Interventions: Other: Diagnostic P-V-loops and MRI
- HFpEF no servere diastolic dysfuntion: LV-EF > 50%, no echocardiographic criteria for diastolic dysfunction, NYHA=>2, Diagnostic P-V-loops and MRI
  Interventions: Other: Diagnostic P-V-loops and MRI
- No HF or diastolic dysfunction: LV-EF > 50%, no diastolic dysfunction, no heart failure, Diagnostic P-V-loops and MRI
  Interventions: Other: Diagnostic P-V-loops and MRI

INTERVENTIONS:
Other: Diagnostic P-V-loops and MRI — Invasive assessment of P-V-loops during catheterization for suspected CAD Magnetic resonance Imaging for assessment of myocardial fibrosis and biventricular function

SUMMARY:
StiffMAP-HFpEF trial is an investigator initiated, observational, single-center study that will evaluate whether fibrosis quantification by cardiac MRI correlates with left and right ventricular stiffness derived from pressure-volume analysis, aiming to clarify if cardiac MRI is a valid, non-invasive method to assess diastolic function in patients with Heart Failure with preserved ejection fraction.

DETAILED DESCRIPTION:
Heart Failure with preserved ejection fraction (HFpEF) and diastolic dysfunction is a growing medical challenge. To date almost every second patient with heart failure has a preserved ejection fraction and recent data show that outcomes in these patients are as bad as in those with reduced ejection fraction. In clinical routine the diagnosis of HFpEF is complicated by indirect assessment of diastolic function. Mechanistically the diastolic dysfunction is among others believed to be caused by the development of diffuse myocardial fibrosis with an increase of extracellular matrix.

Direct assessment of the intrinsic diastolic function and stiffness of the ventricle can be obtained by pressure-volume-curve tracings through a conductance catheter. Although this offers the benefit of assessing load-dependent and load-independent parameters of diastolic function as well as information on contractility and ventricular-arterial coupling, the use of this technique is limited by its invasiveness in daily care.

Newer MRI techniques have made it possible to quantify not only local fibrosis but also diffuse fibrosis (i.e. T1-Mapping) and determine extracellular volumes.

Moreover, the role of right ventricular function is in HFpEF is not well defined.

Aim of the current study is therefore to evaluate the role of MRI in assessing cardiac fibrosis in the context of impaired LV diastolic function in HFpEF patients, as well as to evaluate the role of systolic and diastolic right ventricular functional impairment in this patient cohort.

ELIGIBILITY:
Inclusion Criteria:

* LV-EF > 50%
* Indication for invasive cardiac catheterization

Exclusion Criteria:

* know CAD or CAD in Angiography (stenoses > 50%)
* acute coronary syndromes
* Cerebral ischemia within the last year
* contraindications for MRI
* more than mild valvular disease
* Constrictive pericarditis, restrictive Cardiomyopathy, pericardial effusion
* pregnancy
* enrolment in other study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Recruitment of consequtive patients from our general cardiology clinic that present with signs of heart failure or suspected CAD with indication for invasive assessment and fullfill eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2014-09; Primary Completion 2016-05 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Correlation of extracellular volume (MRI) and myocardial stiffness (p-v-loops) | Baseline

SECONDARY OUTCOMES:
LV stiffness constant (ß) between groups | Baseline
Time constant of LV-relaxation (Ƭ) between groups | Baseline
Change in endiastolic pressure volume relation (EDPVR) under excercise between groups | Baseline
Right Ventricular Endsystolic Elastance Slope | Baseline
Right Ventricular Endsystolic Stiffness Constant | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Lurz, PhD, Principal Investigator — University Heart Center Leipzig
Locations (1):
- Heart Center of the University Leipzig, Leipzig, Germany

REFERENCES:
- [Background] Owan TE, Hodge DO, Herges RM, Jacobsen SJ, Roger VL, Redfield MM. Trends in prevalence and outcome of heart failure with preserved ejection fraction. N Engl J Med. 2006 Jul 20;355(3):251-9. doi: 10.1056/NEJMoa052256. PMID 16855265
- [Background] Bhatia RS, Tu JV, Lee DS, Austin PC, Fang J, Haouzi A, Gong Y, Liu PP. Outcome of heart failure with preserved ejection fraction in a population-based study. N Engl J Med. 2006 Jul 20;355(3):260-9. doi: 10.1056/NEJMoa051530. PMID 16855266
- [Background] Burkhoff D, van der Velde E, Kass D, Baan J, Maughan WL, Sagawa K. Accuracy of volume measurement by conductance catheter in isolated, ejecting canine hearts. Circulation. 1985 Aug;72(2):440-7. doi: 10.1161/01.cir.72.2.440. PMID 4006150
- [Background] Westermann D, Kasner M, Steendijk P, Spillmann F, Riad A, Weitmann K, Hoffmann W, Poller W, Pauschinger M, Schultheiss HP, Tschope C. Role of left ventricular stiffness in heart failure with normal ejection fraction. Circulation. 2008 Apr 22;117(16):2051-60. doi: 10.1161/CIRCULATIONAHA.107.716886. Epub 2008 Apr 14. PMID 18413502
- [Background] Sibley CT, Noureldin RA, Gai N, Nacif MS, Liu S, Turkbey EB, Mudd JO, van der Geest RJ, Lima JA, Halushka MK, Bluemke DA. T1 Mapping in cardiomyopathy at cardiac MR: comparison with endomyocardial biopsy. Radiology. 2012 Dec;265(3):724-32. doi: 10.1148/radiol.12112721. Epub 2012 Oct 22. PMID 23091172
- [Derived] von Roeder M, Kowallick JT, Rommel KP, Blazek S, Besler C, Fengler K, Lotz J, Hasenfuss G, Lucke C, Gutberlet M, Thiele H, Schuster A, Lurz P. Right atrial-right ventricular coupling in heart failure with preserved ejection fraction. Clin Res Cardiol. 2020 Jan;109(1):54-66. doi: 10.1007/s00392-019-01484-0. Epub 2019 May 3. PMID 31053957
- [Derived] Rommel KP, von Roeder M, Oberueck C, Latuscynski K, Besler C, Blazek S, Stiermaier T, Fengler K, Adams V, Sandri M, Linke A, Schuler G, Thiele H, Lurz P. Load-Independent Systolic and Diastolic Right Ventricular Function in Heart Failure With Preserved Ejection Fraction as Assessed by Resting and Handgrip Exercise Pressure-Volume Loops. Circ Heart Fail. 2018 Feb;11(2):e004121. doi: 10.1161/CIRCHEARTFAILURE.117.004121. PMID 29449367
- [Derived] von Roeder M, Rommel KP, Kowallick JT, Blazek S, Besler C, Fengler K, Lotz J, Hasenfuss G, Lucke C, Gutberlet M, Schuler G, Schuster A, Lurz P. Influence of Left Atrial Function on Exercise Capacity and Left Ventricular Function in Patients With Heart Failure and Preserved Ejection Fraction. Circ Cardiovasc Imaging. 2017 Apr;10(4):e005467. doi: 10.1161/CIRCIMAGING.116.005467. PMID 28360259
- [Derived] Rommel KP, von Roeder M, Latuscynski K, Oberueck C, Blazek S, Fengler K, Besler C, Sandri M, Lucke C, Gutberlet M, Linke A, Schuler G, Lurz P. Extracellular Volume Fraction for Characterization of Patients With Heart Failure and Preserved Ejection Fraction. J Am Coll Cardiol. 2016 Apr 19;67(15):1815-1825. doi: 10.1016/j.jacc.2016.02.018. PMID 27081022